CLINICAL TRIAL: NCT05861440
Title: Application of Ultrasound Shear Wave Elastography on the Adjunct Corticosteroid Therapy on Tuberculous Lymphadenitis: a Randomized Control Trial
Brief Title: Applying Shear Wave Elastography for Adjunct Steroid on Tuberculous Lymphadenitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202301222MINA
Record Dates: First submitted 2023-05-07; First posted 2023-05-16 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-04

CONDITIONS: Tuberculous Lymphadenitis
Keywords: tuberculous lymphadenitis, paradoxical upgrading reaction
MeSH Terms: conditions — Tuberculosis, Lymph Node | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjunct corticosteroid and standard anti-tuberculosis agent (Experimental): Prednisolone dosing and duration per study protocol
  Interventions: Drug: Prednisolone; Drug: standard anti-tuberculosis agents
- Standard of care with standard anti-tuberculosis agent (Active Comparator): standard anti-tuberculosis agent
  Interventions: Drug: standard anti-tuberculosis agents

INTERVENTIONS:
Drug: Prednisolone — adjunct steroid per study protocol
  Arms: Adjunct corticosteroid and standard anti-tuberculosis agent
Drug: standard anti-tuberculosis agents — standard anti-tuberculosis agents

SUMMARY:
1. To prospectively collect the radiologic data from the initial phase till the post-treatment phase of tuberculous lymphadenitis.
2. To prospectively investigate the benefits of corticosteroid on reduction of paradoxical upgrading reaction in patients with tuberculous lymphadenitis based on the results of shear wave elastography.
3. To investigate the potential biomarker of host immunity in response to tuberculosis and predict the development of paradoxical upgrading reaction.

DETAILED DESCRIPTION:
Tuberculosis remained one of the top ten leading cause of death worldwide. There were more than 10 million new diagnoses per year, and up to 1.2 million deaths caused by tuberculosis. Extra-pulmonary tuberculosis is defined as infection outside the lung. Tuberculous lymphadenitis is the most common site of extra-pulmonary tuberculosis, constituting around 30-50% of all cases. A unique manifestation with worsening of symptoms, called paradoxical upgrading reaction (PUR), may develop in 20-50% of patients with tuberculous lymphadenitis during the therapy. Common presentations of the PUR include swollen lymphadenitis with pain or rupture with pus. Patients may fail to complete the treatment and jeopardize the development of drug-resistant pathogen. Limited studies investigated the risk factors associated with the PUR. In our prior study, ultrasound shear wave elastography offers quantified values as the objective parameters to successfully predict the occurrence of PUR. In this study, we aim to investigate the effect of corticosteroid as an adjunct therapy to reduce the PUR from happening in patients with tuberculous lymphadenitis.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed of tuberculous lymphadenitis.
* The diagnosis of tuberculous lymphadenitis must qualify any of the following criteria:

  1. microbiological evidence (culture or nucleic acid amplification test)
  2. histology specimen featuring caseating granulomatous inflammation with acid-fast bacilli on smear, or clinical response to anti-tuberculosis therapy.

Exclusion Criteria:

* Participants with age < 18 years
* Diagnoses based on histologic report turned out to be non-tuberculosis mycobacterial infection
* The tuberculous lymphadenitis involved was surgically removed, without available target to be monitored
* Participant under systemic (oral or parenteral) steroid therapy.
* Participant with active hepatitis B virus infection
* Participant reluctant to be enrolled in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
reduction rate of paradoxical upgrading reaction | up to 9 months
  decreased in occurrence of unpredicted paradoxical reaction

SECONDARY OUTCOMES:
hospital-anxiety scale | up to 9 months
  The objective measurement of anxiety status by scoring, ranging from 0-21. Score with the higher value suggest more severe anxiety.
hospital- depression scale | up to 9 months
  The objective measurement of depression status by scoring, ranging from 0-21. Score with the higher value suggest more severe depression.
tuberculosis relapse rate | up to 24 months
  recurrence of tuberculosis infection
treatment duration | up to 9 months
  total duration of anti-tuberculosis drug
adverse events during corticosteroid therapy | up to 9 months
  any side effects of drugs related or associated with corticosteroid
paradoxical upgrading reaction rate in low elasticity group | up to 9 months
  the occurrence of paradoxical reaction in non-steroid using group

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Lin Chen, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen YL, Kuo YW, Wu HD, Wang JY, Wang HC. The application of ultrasound shear wave elastography in the prediction of paradoxical upgrading reaction in tuberculous lymphadenitis. a pilot study. J Formos Med Assoc. 2022 Sep;121(9):1696-1704. doi: 10.1016/j.jfma.2021.12.002. Epub 2021 Dec 23. PMID 34953644
- [Background] Kuo YW, Chen YL, Wu HD, Chien YC, Huang CK, Wang HC. Application of transthoracic shear-wave ultrasound elastography in lung lesions. Eur Respir J. 2021 Mar 25;57(3):2002347. doi: 10.1183/13993003.02347-2020. Print 2021 Mar. PMID 33033150